CLINICAL TRIAL: NCT06759740
Title: An Exploratory Study of 68Ga-DOTA-SEMA in Preoperative Precise Imaging of Patients with Glucagon-Like Peptide-1 Receptor (GLP1R) Positive Insulinomas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator did not plan to carry out this study and voluntarily withdrew it
Sponsor: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Xie Yang, Director, The Affiliated Hospital Of Southwest Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AHSWMU-2024-072
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Hypoglycaemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Radiation: 68Ga-DOTA-SEMA

INTERVENTIONS:
Radiation: 68Ga-DOTA-SEMA — 68Ga-DOTA-SEMA is GLP1R imaging agent

SUMMARY:
Traditional imaging techniques for insulinomas have a low detection rate. This study aims to evaluate the safety, internal radiation dosimetry, and targeted imaging capability of the novel GLP1R imaging agent, 68Ga-DOTA-SEMA, in patients with GLP1R-positive insulinomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are capable of understanding and voluntarily signing an approved informed consent form (ICF).
2. Age ≥ 18 years.
3. Normal renal function (serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 50 mL/min, and estimated glomerular filtration rate (eGFR) > 80 mL/min/1.73 m²).
4. Recurrent hypoglycemia with biochemically confirmed endogenous hyperinsulinemic hypoglycemia (at least 3 episodes of biochemically confirmed endogenous hyperinsulinemic hypoglycemia within the past 3 months, each with detailed blood glucose monitoring records and symptom descriptions confirming endogenous hyperinsulinemia as the cause).
5. Negative for sulfonylurea drugs and insulin autoantibodies.
6. ECOG performance status ≤ 2, able to tolerate the examination.
7. All other toxicities must be ≤ NCI-CTCAE v5.0 Grade 0 or 1.

Exclusion Criteria:

1. History of allergy or hypersensitivity to the components or excipients of the investigational drug.
2. Claustrophobia or inability to tolerate imaging procedures for other reasons.
3. Clinically significant active infection as determined by the investigator.
4. History or current presence of uncontrolled primary or metastatic brain tumors.
5. Serious and/or uncontrolled and/or unstable conditions that may affect the study as judged by the investigator, including but not limited to:

   1. Poorly controlled diabetes.
   2. Congestive heart failure.
   3. Myocardial infarction within the past 12 months.
   4. Uncontrolled and unstable hypertension.
   5. Chronic kidney disease or liver disease.
   6. Severe pulmonary diseases.
6. Poor compliance and inability to complete study procedures as expected.
7. Any other conditions that the investigator considers unsuitable for participation in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radiation dose to major organs and tumors | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan, China